CLINICAL TRIAL: NCT00366392
Title: Project Magnify - A Comparison of Two Strategies (Large Print Versus Optical Aids) for Helping Visually Impaired Students Improve Reading Abilities
Brief Title: Project Magnify - A Comparison of Two Strategies to Improve Reading Ability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: South Carolina School for the Deaf and the Blind (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEI-05-001
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2006-07

CONDITIONS: Vision, Low
Keywords: Low Vision; Optical Aids
MeSH Terms: conditions — Vision, Low

INTERVENTIONS:
Device: Optical Aids

SUMMARY:
The purpose of Project Magnify is to determine which of the two current strategies (large print versus optical aids) for helping visually impaired students improve their reading abilities works better. Our hypothesis is that optical aids work better than providing the student with large print materials. Since large print materials are of one size only, and the level of visual impairments among students varies greatly, it seems apparent that large print materials will work well for some students, but not for all. An optical aid designed for each individual student's level of impairment seems to hold more promise in helping each student reach their maximum level of performance. Although Project Magnify is designed to increase reading abilities, it is expected that students will also develop greater independence and confidence in home and community activities that require the use of vision.

DETAILED DESCRIPTION:
The purpose of Project Magnify is to determine which of the two current strategies (large print versus optical aids) for helping visually impaired students improve their reading abilities works better. Our hypothesis is that optical aids work better than providing the student with large print materials. Since large print materials are of one size only, and the level of visual impairments among students varies greatly, it seems apparent that large print materials will work well for some students, but not for all. An optical aid designed for each individual student's level of impairment seems to hold more promise in helping each student reach their maximum level of performance. Although Project Magnify is designed to increase reading abilities, it is expected that students will also develop greater independence and confidence in home and community activities that require the use of vision.

Students with low vision are frequently given large print books to read. Large print does give many students the opportunity to access information in textbooks. However, there are several limitations to this strategy. First, the student only has access to the print that has been enlarged for him. And large print material is of only one size, while student's level of vision impairment varies greatly. So the large print may be fine for one visually impaired student, but significantly too small for another, and way too big for yet a third. When large print is a child's only option for accessing print, he struggles to copy notes off the board, find the right bus in the bus line and correctly measure the chemicals in the science laboratory experiment. Additionally, the difficulties and costs related to enlarging colored pictures, graphs and charts result in second rate productions of graphics; thereby, hindering comprehension of critical information. Furthermore, the cost of large print books is exorbitant. According to Jill Ischinger the Director of the South Carolina Instructional Resource Center (personal communication), IRC, the cost of providing a set of books to students each year is approximately $2,237. Finally, students who choose to further their education beyond high school are severely limited with reading options. Unlike primary and secondary school where the Department of Education purchased the textbooks and the books were generally available in large print, college students frequently lack the resources to pay for the costly, rare books.

Moreover, previous studies have found that the reading rates of large print readers are not commensurate with their regular print readers. With the current pressure of high stakes testing and greater achievement, readers with visual impairments are at an increased risk of falling further behind in school.

Project Magnify is modeled after a successful study sponsored by Vanderbilt University in Tennessee: Providing Access to the Visual Environment (PAVE). PAVE provides comprehensive low vision services to school aged children throughout the state of Tennessee. The services provided by PAVE include clinical low vision evaluations and instruction in the use of the low vision aids. When PAVE was initiated, Corn, Wall and Bell researched the reading rates of students with low vision reading with optical aids to the reading rates of non-visually impaired students. The study showed that while students with visual impairments continue to lag behind their peers in reading rates optical aids significantly reduce the disparity (1999). Our study is designed to replicate a portion of this pioneer study and expand upon it by comparing the two dominant methods of helping visually impaired students improve their reading skills: large print versus optical aids.

Whereas PAVE compared the reading rates of optical aid users to their sighted peers, Project Magnify seeks to determine the benefits of optical aids as compared to large print. In our study design, the students using large print alone will be the control group. Students in the experimental group will use an optical aid prescribed specifically for their use. The main outcome measures are the reading tests that are conducted before and after the twelve month reading treatments. The differences in the before and after reading rates are compared to determine statistical significance. Since the reading rates are on a normal numerical scale, parametric statistics can be used to compare the different reading rates. A Students T-test will allow us to compare the differences in reading rates for the two groups of visually impaired students. To conduct this study, twenty students currently served by the South Carolina School for the Deaf and the Blind Division of Outreach Services (SCSDB) will be referred for inclusion in the study. The reading levels of all of the students will be assessed with a formal reading assessment. Students will then be randomly assigned to two groups. The large print readers in the control group will receive instruction as currently indicated on their Individual Education Plans (IEPs). Students in the second group will travel to the Feldberg Center in Charleston for a clinical low vision evaluation. Furthermore, these students will receive monthly instruction in the use of the low vision aids throughout the duration of the study. At the study's close, reading levels of the students in both groups will be assessed. The change in reading rates of the students will be compared to determine whether a significance difference exists between optical aids and large print.

ELIGIBILITY:
Inclusion Criteria:

* visually impaired with a permanent reduction of visual acuity in both eyes equal to or less than 20/70
* enrolled in one of the South Carolina school districts served by the South Carolina School for the Deaf and Blind (SCSDB) outreach Teachers of the Visually Impaired (VI)
* previously taught using large print materials without optical aids, or magnifiers
* 5 to 17 years of age

Exclusion Criteria:

* none

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2005-05; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Morse, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Feldberg Center for Vision Rehabilitation, Medical University of South Carolina, Charleston, South Carolina, United States